CLINICAL TRIAL: NCT03858387
Title: Pharmacokinetics/Pharmacodynamics and Clinical Outcomes of β-lactams in Critically Ill Patients
Brief Title: PK/PD and Clinial Outcomes of Beta-lactams in ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sutep Jaruratanasirikul, Department of Medicine, Faculty of Medicine, Prince of Songkla University, Prince of Songkla University
Other Study IDs: B-lactams-ICU-61061141
Record Dates: First submitted 2019-02-24; First posted 2019-02-28 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Critical Illness; Bacterial Infections
Keywords: pharmacokinetics; pharmacodynamics; meropenem; imipenem
MeSH Terms: conditions — Critical Illness; Bacterial Infections | interventions — Meropenem; Imipenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Meropenem: Critically ill patients who require meropenem therapy
  Interventions: Drug: Meropenem
- Imipenem: Critically ill patients who require imipenem therapy
  Interventions: Drug: Imipenem

INTERVENTIONS:
Drug: Meropenem — This group is composed of 52 critically ill patients, meropenem dosage is chosen by the intensivist in charge of the case.
  Blood sampling: 5 blood samples (3 mL) were obtained from a heparinized intravascular catheter by direct venipuncture at the following time: before (time 0) and during 0-0.5 h, 0.5-2.5 h, 2.5-4 h, 4-8 h or 4-12 after meropenem administration.
  Groups: Meropenem
Drug: Imipenem — This group is composed of 50 critically ill patients, imipenem dosage is chosen by the intensivist in charge of the case.
  Blood sampling: 5 blood samples (3 mL) were obtained from a heparinized intravascular catheter by direct venipuncture at the following time: before (time 0) and during 0-0.5 h, 0.5-2 h, 2-4 h, 4-6 h or 4-12 after imipenem administration.
  Other Names: Imipenem/cilastatin
  Groups: Imipenem

SUMMARY:
Meropenem and imipenem are broad-spectrum carbapenem antibiotic and are frequently prescribed in critically ill patients with severe infections. These patients show several pathophysiological changes that may alter the carbapenem pharmacokinetic (PK) normally found in other populations. Although the PK of carbapenems has been widely studied, most studies have been conducted on small populations, and clinical outcome data are sparse. Therefore, the aims of this study are (i) describe the population pharmacokinetic parameters of meropenem and imipenem in critically ill subject (ii) evaluate the pharmacodynamic of meropenem and imipenem as a predictor of clinical treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* severely ill patient who admitted to medical or surgical intensive care unit who require a treatment with meropenem or imipenem antibiotic

Exclusion Criteria:

* severe renal impairment and require renal replacement therapy
* APACHE II score >30
* History of hypersensitivity to carbapenems
* Pregnancy or breast-feeding female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Population pharmacokinetic parameters of meropenem and imipenem | 24-48 hours after treatment
%fT>MIC of meropenem and imipenem | 24-48 hours after treatment
  the percentage of time which the free drug concentration remains above the minimum inbibitory concentration (%fT>MIC)

SECONDARY OUTCOMES:
The relationship between %fT>MIC and clinical cure | Day 3-7 after treatment and end of therapy (7-14)
  Clinical cure: disappearance of all signs and symptoms related to the infection, such that no additional antibacterial therapy, drainage, or surgical procedure was required.
The relationship between %fT>MIC and microbiological cure | Day 3-7 after treatment and end of therapy (7-14)
  Success is eradication (absence of the baseline pathogen in a specimen appropriately obtained from the original site of infection) or presumed eradication (absence of material to culture in a subject who was assessed as a clinical cure).
The relationship between %fT>MIC and mortality | during hospital stay and at day 28
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sutep Jaruratanasirikul, M.D., Principal Investigator — Faculty of Medicine, Prince of Songkla University, Thailand
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Thailand, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Derived] Jaruratanasirikul S, Boonpeng A, Nawakitrangsan M, Samaeng M. NONMEM population pharmacokinetics and Monte Carlo dosing simulations of imipenem in critically ill patients with life-threatening severe infections during support with or without extracorporeal membrane oxygenation in an intensive care unit. Pharmacotherapy. 2021 Jul;41(7):572-597. doi: 10.1002/phar.2597. Epub 2021 Jun 18. PMID 34080708